CLINICAL TRIAL: NCT05596604
Title: "Awareness, Preconception, and Fear of Epidural Analgesia Among Childbearing Women in Saudi Arabia."
Status: Completed | Type: Observational
Sponsor: King Khalid University Hospital (Other)
Collaborators: King Saud University (Other)
Responsible Party: Principal Investigator, Abdulrhman Alshihri, general practitioner, King Khalid University Hospital
Other Study IDs: 4361020
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Assess Women Awareness and Fear About EDA for Labor
Keywords: Awareness, preconception, fear, epidural analgesia, labor pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey- no intervention — survey- no intervention

SUMMARY:
The aim of our study is to measure the level of awareness, preconceptions, and level of fear regarding epidural analgesia among childbearing women in KKUH in Riyadh.

DETAILED DESCRIPTION:
This research was designed as a hospital-based observational cross-sectional study conducted at King Khalid University Hospital, using a self-administered questionnaire based on previous research.22-24-26 approved by the Institutional Review Board at King Saud University, College of Medicine, Riyadh, Saudi Arabia on 08.August.2022 Ref. No. 22/0592/IRB. The sample included pregnant women attending an obstetrical clinic for routine antenatal follow-up, and the data collection was conducted during the month of August 2022. The questionnaire included five parts (sociodemographic, preconception, awareness, fear, and desirability). a total of 26 questions with multiple-choice answers. The sample size was determined using the Comrey and Lee criterion Comrey and Lee (1992) stated that a 200-sample size is acceptable. The questionnaire was completed by 202 participants who met the inclusion criteria that is being a pregnant woman and completing the survey, and the exclusion criteria were non-pregnant women and an incomplete survey. The data collectors made it clear to the participants that taking part in the study was completely optional, and the participants signed anonymous consent forms.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman
* completing the survey

Exclusion Criteria:

* non-pregnant women
* incomplete survey

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: included pregnant women attending an obstetrical clinic for routine antenatal follow-up
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Awareness | month
  assess awareness among participants

CONTACTS AND LOCATIONS:
Locations (1):
- King Khalid Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
we are not planning to share data